CLINICAL TRIAL: NCT06900855
Title: Prevalence, Causes and Demographic Profile of Patients Seeking a Visual Impairment Certificate
Brief Title: Patients Seeking a Visual Impairment Certificate
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madona Gerges Boles, resident at Ophthalmology department, Assiut University
Other Study IDs: visual impairment certificate
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Demographic Profiles; Impairment Certificates; Visual Impairment
Keywords: visual impairment; demographic profiles; visual impairment certificates
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Seeking Visual Impairment Certificates at Assiut Ophthalmology Hospital: The study population consists of patients requesting visual impairment certificates at Assiut Ophthalmology Hospital, who have undergone all required investigations, including visual field testing, OCT macula imaging, VEP, ERG, ultrasound, and fundus photography. Eligible participants are those fulfilling WHO's definition of blindness, defined as having best-corrected distance visual acuity (BCVA) of 3/60 or less in the better eye or a visual field restricted to 10° or less in the widest diameter of vision. Excluded are patients unwilling to participate or with incomplete/missing investigations. A calculated sample size of 383 cases ensures statistical reliability. Demographic and clinical data such as age, sex, occupation, socioeconomic status, marital status, education level, and associated systemic conditions are collected alongside comprehensive eye examinations.

SUMMARY:
This study investigates the prevalence, causes, and demographic characteristics of patients seeking visual impairment certificates at Assiut Ophthalmology Hospital. Using a prospective cross-sectional design, it aims to identify the magnitude and nature of visual impairment in this population by analyzing clinical data, performing comprehensive eye examinations, and utilizing advanced diagnostic tools.

DETAILED DESCRIPTION:
The study is designed to explore the prevalence, underlying causes, and demographic profiles of patients requesting visual impairment certificates at Assiut Ophthalmology Hospital. It employs a prospective cross-sectional approach, recruiting patients from ophthalmology outpatient clinics who meet the World Health Organization's (WHO) definition of blindness. Blindness is defined as having best-corrected distance visual acuity (BCVA) of 3/60 or less in the better eye or a visual field restricted to 10° or less in the widest diameter of vision.

Eligible participants undergo comprehensive eye examinations, including visual acuity measurement using Snellen charts, slit-lamp biomicroscopy, dilated fundus examination, and automated perimetry for visual field assessment. Advanced investigations such as OCT macula imaging, VEP (visual evoked potential), ERG (electroretinography), ultrasound, and fundus photography are performed to identify the causes of visual impairment. Demographic data-such as age, sex, marital status, occupation, socioeconomic status, education level-and systemic medical history are collected to assess contributing factors.

The sample size was calculated using Epi-info software with a confidence level of 95% and confidence limits of 5%, estimating a minimum of 383 cases. By analyzing clinical findings alongside demographic characteristics, the study aims to provide valuable insights into the magnitude and nature of visual impairment in this specific population. This information could help inform public health strategies and improve services for visually impaired individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients requesting visual impairment certificate at Assiut ophthalmology hospital having all investigations Visual field, OCT macula, VEP, ERG, US, Fundus photography Werepatients who fulfilled WHO's definition of blindness. The blind patients according to WHO's,were defined as patients having best corrected distance visual acuity (BCVA) of 3/60 or less in the better eye or a visual field restricted to 10 or less in the widest diameter of vision.

Exclusion Criteria:

* Patients unwilling to participate in the study Incomplete or missing investigations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants undergo comprehensive eye examinations, including visual acuity measurement using Snellen charts, slit-lamp biomicroscopy, dilated fundus examination, and automated perimetry for visual field assessment. Advanced investigations such as OCT macula imaging, VEP (visual evoked potential), ERG (electroretinography), ultrasound, and fundus photography are performed to identify the causes of visual impairment. Demographic data-such as age, sex, marital status, occupation, socioeconomic status, education level-and systemic medical history are collected to assess contributing factors.
Sampling Method: Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
BCVA | 1 month
  BCVA of 3/60 or less in the better eye visual field restricted to 10 or less in the widest diameter of vision.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Journal of Research in Medical Sciences Priya M et al. Int J Res Med Sci. 2023 Aug
- [Background] Bourne et al. (2013). Prevalence and causes of vision loss in high-income countries: a review. Lancet Global Health